CLINICAL TRIAL: NCT04552067
Title: Generic and Branded Enoxaparin Bioequivalence: a Randomized Study in Acute Coronary Syndrome Patients With an In-vitro Thrombin Generation Testing Comparison
Brief Title: Enoxaparin Bioequivalence Study in Acute Coronary Syndrome Patients
Acronym: Enoxaparine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Monastir (Other)
Collaborators: University Hospital Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Head of departement, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Enoxaparine
Record Dates: First submitted 2020-02-20; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Acute Coronary Syndrome
Keywords: enoxaparin; Lovenox; ani-Xa; acute coronary syndrome; Enoxa
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LOVENOX (Other): patients are given a curative dose of Enoxaparin (LOVENOX)
  Interventions: Drug: Lovenox
- Enoxamed (Active Comparator): patients are given a curative dose of Enoxaparin (ENOXA)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Lovenox — patients given curative dose of Lovenox
  Arms: LOVENOX
Drug: Enoxaparin — patients given curative dose of Enoxa
  Other Names: Enoxamed
  Arms: Enoxamed

SUMMARY:
Because of their anti-Xa and ease of administration activity, the Low molecular weight heparin represent an attractive alternative to the unfractionated heparin. Several clinical trials have demonstrated that Low molecular weight heparin was more effective than Unfractionated heparin without increasing bleeding complications. Enoxaparin has been the most studied. Its use is recommended.

Demonstrate that Enoxa® is comparable to that of Lovenox® in the anti-Xa activity action.

DETAILED DESCRIPTION:
Single-center randomized controlled trial, single-blind, including patient with an acute coronary syndrome confirmed, to measure the anti-Xa activity between H0 and H4.the study was done on two groups ; ENOXA® group : In this case the patient is given an injection of enoxaparin ( ENOXA® ; UNIMED Laboratories) intravenously. Curative dose (100 IU/10 kg).

Control group ( LOVENOX ® ):

In this case the patient receives LOVENOX intravenous injection curative dose of 100 kg IU/10 .

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 year old
* With an acute coronary syndrome confirmed

Exclusion Criteria:

* Age less than 18 years
* Persistent ST segment elevation
* Contre indication of enoxaparin and heparin in general.
* Patient participating in another study,
* Pregnant or nursing women
* patients taking an anticoagulant in the last three months,
* Patients with coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
anti Xa activity (UI/ml) | 4 hours
  Compare the Anticoagulant Activity (measured in a UI per ml in a reference laboratory) of Two Formulations of Enoxaparin [ENOXA ® Versus LOVENOX ®], Conducted on Two Parallel Groups of Patients Admitted to Emergency for Acute Coronary Syndrome

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 30 days
  All major cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University hospital of Monastir
Locations (1):
- Emergency Department of University Hospital of Monastir, Monastir, Tunisia

REFERENCES:
- See also: official website — http://www.urgencemonastir.com